CLINICAL TRIAL: NCT07358221
Title: Impact of Different Cardioplegia Solutions on Extracellular Vesicles-derived miRNAs, Complement System, and Neutrophil Extracellular Traps (NETs) as Indicators of Myocardial Injury During Coronary Artery Bypass Surgery
Brief Title: Impact of Different Cardioplegia Solutions on Indicators of Myocardial Injury During Coronary Surgery
Acronym: Cardioplegia2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Principal Investigator, Mohammad Bashar Izzat, Professor, Damascus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Cardioplegia2
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Bypass Grafting (CABG) Surgery; Myocardial Protection
Keywords: coronary surgery; cardioplegia; complement activation; myocardial injury

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- St. Thomas' cardioplegia (Active Comparator): Intervention: Patients in this group will be managed with St. Thomas' cold crystalloid cardioplegia solution during surgery
  Interventions: Procedure: The intervention is the use of a specific cardioplegia solution for myocardial protection
- Calafiore cardioplegia (Active Comparator): Patients in this group will be managed with Calafiore warm blood intermittent cardioplegia solution during surgery
  Interventions: Procedure: The intervention is the use of a specific cardioplegia solution for myocardial protection
- del Nido cardioplegia (Active Comparator): Patients in this group will be managed with del Nido cold blood intermittent cardioplegia solution during surgery
  Interventions: Procedure: The intervention is the use of a specific cardioplegia solution for myocardial protection

INTERVENTIONS:
Procedure: The intervention is the use of a specific cardioplegia solution for myocardial protection — Three different solutions will be used for myocardial protection in this study, and will be compared using markers of myocardial injury

SUMMARY:
The aim of the present study is to investigate intra-operative changes in markers of myocardial injury during ischemia and reperfusion, comparing three methods of myocardial protection; St. Thomas' cold crystalloid cardioplegia, Calafiore warm blood cardioplegia, or modified del Nido cold blood cardioplegia in routine coronary artery bypass grafting procedures.

DETAILED DESCRIPTION:
Thirty consecutive patients undergoing elective primary coronary artery bypass grafting will be enrolled in this study. Patients were excluded from this study if they had suffered from previous myocardial infarction, had reduced ejection fraction or were undergoing combined or repeated surgery. Patients will be randomly assigned to undergo surgery using one of three methods for myocardial protection: Group 1: St. Thomas' cold crystalloid cardioplegia (consisting of 750 ml of normal saline solution, 110 - 147 mmol/L of sodium chloride, . 16 - 20 mmol/L of potassium chloride, 16-32 mmol/L of magnesium chloride, 1.2-2.4 mmol/L of Calcium Chloride, 10 mmol/L of Sodium Bicarbonate). This solution will be administered as a 1-liter bolus at 3-4 degrees C following application of the aortic cross-clamp, and repeated as a 500 ml bolus if cross-clamp time extended beyond 30 minutes. Group 2: Calafiore intermittent antegrade warm blood cardioplegia (consisting of normothermic pump blood, potassium chloride 2 mEq/ml and magnesium sulfate 50%). This cardioplegic solution will be administered at 37 degrees C following application of the aortic cross-clamp and repeated after completion of each distal coronary anastomosis. • Group 3: Modified del Nido intermittent antegrade cold blood cardioplegic solution (consisting of 750 ml of lactated Ringer solution, 200 ml of pump blood, 13 ml of sodium bicarbonate 8.4%, 16 ml of mannitol 20%, 4 ml of magnesium sulfate 50%, 13 ml of lidocaine 2% and 13 ml of potassium chloride 2 mEq/ml). This solution will be administered as a 1-liter bolus at 3-4 degrees C following application of the aortic cross-clamp, and repeated as a 500 ml bolus if cross-clamp time extended beyond 60 minutes.

Collection of blood samples and myocardial biopsies:

Peripheral blood samples will be collected immediately prior to surgery, 15 minutes after removal of cross-clamp, and at 6 hours and 24 hours postoperatively. Myocardial biopsies (4-14 mg wet weight) will be taken using a Tru-cut needle from the apex of the left ventricle in every patient as follows: Biopsy 1: "Resting specimen", immediately after beginning of extracorporeal circulation. Biopsy 2: "Ischemic specimen", 30 minutes after application of the aortic cross-clamp. Biopsy 3: "Reperfusion specimen", 20 minutes following the removal of aortic cross-clamp. Each specimen will be immediately snap-frozen in liquid nitrogen (-185 degrees C) until processing.

Extracellular vesicles-derived miRNA (miR-499, miR-208b, miR-133a, EV-miR-1) will be measured, and release kinetics of EV-miRNAs will be determined and compared between the three groups, including correlation between EV-miRNA and cross-clamp time.

Complement system activation (sC5b-9, C5a, C3a) will be determined and compared between the three groups, including whether blood cardioplegia reduces complement activation and the relation between cardioplegia temperature and complement activation.

Neutrophil extracellular Traps (dsDNA) will be determined and compared between the three groups, including the effect of hypothermia on NETs formation.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing elective primary coronary artery bypass grafting will be enrolled in this study.

Exclusion Criteria:

* Patients will be excluded from this study if they had suffered from previous myocardial infarction, had reduced ejection fraction or were undergoing combined or repeated surgery

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Changes in extracellular vesicles-derived miRNAs as markers of myocardial injury | From start of surgery and for 24 hours
  Extracellular vesicles-derived miRNA (miR-499, miR-208b, miR-133a, EV-miR-1) will be measured, and release kinetics of EV-miRNAs will be determined and compared between the three groups, including correlation between EV-miRNA and cross-clamp time.
Changes in complement system activation | from start of surgery and for 24 hours
  Complement system activation (sC5b-9, C5a, C3a) will be determined and compared between the three groups, including whether blood cardioplegia reduces complement activation and the relation between cardioplegia temperature and complement activation.
Changes in neutrophil extracellular traps (NETs) | From start of surgery and for 24 hours
  Neutrophil extracellular Traps (dsDNA) will be determined and compared between the three groups, including the effect of hypothermia on NETs formation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad B Izzat, FRCS(CTh), Study Chair — Damascus University School of Medicine
Locations (1):
- Damascus University Cardiac Surgery Hospital, Damascus, Rif-dimashq Governorate, Syria

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded on (figshare) data repository site
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Information will be made available in March 2027 and will be available permanently
Access Criteria: open to all

REFERENCES:
- [Background] Zhou X, Mao A, Wang X, Duan X, Yao Y, Zhang C. Urine and serum microRNA-1 as novel biomarkers for myocardial injury in open-heart surgeries with cardiopulmonary bypass. PLoS One. 2013 Apr 22;8(4):e62245. doi: 10.1371/journal.pone.0062245. Print 2013. PMID 23630629
- [Background] Lai KB, Sanderson JE, Izzat MB, Yu CM. Micro-RNA and mRNA myocardial tissue expression in biopsy specimen from patients with heart failure. Int J Cardiol. 2015 Nov 15;199:79-83. doi: 10.1016/j.ijcard.2015.07.043. Epub 2015 Jul 13. PMID 26188824